CLINICAL TRIAL: NCT06746155
Title: Predictors of Early Relapse During Follow-up of Remitted Major Depression
Brief Title: Predictors of Relapse in Major Depressive Disorder
Acronym: PERFORM-D
Status: Recruiting | Type: Observational
Sponsor: Abraham Nunes (Other)
Collaborators: McMaster University (Other); University of British Columbia (Other); University of Calgary (Other); Ontario Shores Centre for Mental Health Sciences (Other); Queen's University (Other); Nova Scotia Health Authority (Other); University Health Network, Toronto (Other); University of Ottawa (Other); Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor-Investigator, Abraham Nunes, Psychiatrist/Assistant Professor, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Other Study IDs: CAN-BIND-20
Record Dates: First submitted 2024-10-30; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Major Depressive Disorder; Remission; Follow-up; Biomarkers; Relapse; Clinical predictors; Relapse prediction
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Major depressive disorder (MDD) is a common condition involving recurring periods of depression. One of the major challenges faced by people with MDD is that the episodes of depression tend to recur even after they are successfully treated. Currently, it is hard to predict when a depressive episode will recur. Being able to forecast this would help healthcare providers monitor patients and prevent relapse.

The purpose of this study is to monitor features such as clinical symptoms, physical activity, sleep patterns, cognitive functioning and brain activity to help us understand how relapse happens and the mechanisms that cause it. From these different types of data, investigators will build a model that tells us who is more likely to experience a relapse and when the relapse is likely to occur.

This study will be a significant step forward in understanding and managing MDD. Investigator will create a practical tool that will allow healthcare providers to monitor patients more effectively. By identifying early signs of relapse, investigators may be able to intervene promptly to prevent depressive episodes. Finally, our research will help understand the factors that underlie relapse in MDD, which will encourage the development of novel treatment approaches.

DETAILED DESCRIPTION:
This study is a multi-centre prospective naturalistic observational cohort study. Participants will be enrolled and followed for 18 months since enrollment. This study will be conducted across nine Canadian clinical-academic sites (Vancouver, Calgary, Hamilton, Toronto Western Hospital, Toronto-Center for Addiction and Mental Health [CAMH], Kingston, Ottawa, Ontario Shores and Halifax), which are currently enrolling participants for the OPTIMUM-D study (NCT05017311). For the present study, participants will be recruited from each of these sites, focusing on OPTIMUM-D participants who attain broadly-defined remission.

Participants will wear a GENEActiv accelerometer (Activinsights; motion tracker) on the non-dominant wrist for the duration of the study. Participants will rate their depression by completing the Quick Inventory of Depressive Symptoms 16-item Self-Rated Version (QIDS-16SR) and anxiety by completing the Generalized Anxiety Disorder 7-item (GAD-7) at weekly interval throughout the study. Participants will have bi-monthly in-person follow-up assessments to rate their depressive symptom severity using the Montgomery-Asberg depression Rating Scale (MADRS). Speech and Electroencephalography (EEG) will be collected bi-monthly, and at the time of relapse.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients 18 to 70 years of age.
* Meet DSM-V criteria for MDD as determined by the SCID-5.
* In the current or most recent MDE, participant must be responding or responded to a treatment or a combination of treatments for MDD. Patients with remitted MDD who are currently not taking medications will also be accepted.
* Participants must have a MADRS total score ≤14.
* Participant must be willing and able to complete self-reported assessments including sufficient fluency in English.
* Participant must be willing to wear the wrist-worn actigraphic device for the duration of the study.

Exclusion Criteria:

* Bipolar I or Bipolar-II diagnosis (lifetime), schizophrenia, or schizoaffective disorder.
* Elevated risk of suicide, as determined by clinical evaluation.
* Existence of major neurological disorders, head injury (if accompanied by any of [A] loss of consciousness longer than 24 hours, [B] documented evidence of Glasgow Coma Scale <9 at the time of injury, [C] post-traumatic amnesia lasting longer than 24 hours) (43), or other unstable medical conditions.
* The participant presents with any condition which, according to the researcher's judgment, could interfere with the assessments stipulated in the protocol.
* The participant is employed by the researcher, actively involved in the current study or other research overseen by the same researcher, or is a relative of a study employee or the researcher.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who participated in the OPTIMUM-D protocol, and who are currently in remission. Past participants from other CAN-BIND studies who meet current inclusion/exclusion criteria will also be approached for the present study. Other patients with MDD, currently in remission, who attend clinics at each of the study sites will also be considered for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Time-to-relapse | 18 months
  In this study, relapse will be defined as any of the following:
  * MADRS total score equal or greater than 22 for at least 2 consecutive weeks. If the relapse criterion of MADRS total score equal or greater than 22 is met at a study visit (scheduled or unscheduled), an additional visit (i.e., the Relapse Verification visit) will be scheduled 2 weeks later (± 5 days) to verify the relapse.
  * Hospitalization onto an inpatient acute care unit for worsening of depression.
  * Suicidal ideation with intent, or suicidal behavior plus at least one elevated MADRS total score of equal or greater than 22.
  * Change in antidepressant management undertaken for the purpose of managing emergent depressive symptoms.
  * Other factors deemed by clinician to be sufficient to denote relapse (the investigator will be asked to describe clinical rationale in this situation).
  Participants who relapse will continue to be followed in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Undecided